CLINICAL TRIAL: NCT04534426
Title: Influence of Different Topical Arnica and Mucopolysaccharide Polysulfate on Postoperative Pain, Edema and Trismus After Extraction of Impacted Third Molar
Brief Title: Topical Arnica and Mucopolysaccharide Polysulfate on Postoperative Pain, Edema and Trismus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Koray Onur Sanal, Assistant Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Abant Izzet Baysal University; 2018/284 (Other: Clinical Researches and Ethics Committee of Bolu Abant Izzet Baysal University)
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Impacted Third Molar Tooth
Keywords: impacted third molar; oral surgery; edema; trismus; pain; postoperative sequelae
MeSH Terms: conditions — Edema; Trismus; Pain | interventions — Arnicae flos extract; mucopolysaccharide polysulfate; Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Postoperative topical arnica montana cream (Active Comparator): In this arm, Arnica group consisted of 20 patients who were treated with topical arnica in addition to standard therapy (amoxicillin/clavulanic acid 500/125 mg twice a day and diclofenac potassium 50 mg twice a day) after mandibular impacted third molar surgery.
  Interventions: Drug: : Arnica montana
- Postoperative topical mucopolysaccharide polysulfate cream (Active Comparator): In this arm, Mucopolysaccharide polysulfate group consisted of 20 patients who were treated with topical arnica in addition to standard therapy (amoxicillin/clavulanic acid 500/125 mg twice a day and diclofenac potassium 50 mg twice a day) after mandibular impacted third molar surgery.
  Interventions: Drug: Mucopolysaccharide polysulfate
- Control group (Other): In this arm control group consisted of 20 patients who were treated with only standard therapy (amoxicillin/clavulanic acid 500/125 mg twice a day and diclofenac potassium 50 mg twice a day) after mandibular impacted third molar surgery.
  Interventions: Other: Control group

INTERVENTIONS:
Drug: : Arnica montana — In Arnica group, patients were given an unlabelled tube containing cream to be applicated topically on skin surface of masseteric and submandibular region, 2 cm in length cream for each 8 hours, starting immediately after surgery and continued for 10 days
  Other Names: Arnika Krem
  Arms: Postoperative topical arnica montana cream
Drug: Mucopolysaccharide polysulfate — In Arnica group and MPSP group, patients were given an unlabelled tube containing cream to be applicated topically on skin surface of masseteric and submandibular region, 2 cm in length cream for each 8 hours, starting immediately after surgery and continued for 10 days
  Other Names: Hirudoid Fort Krem 445mg/100g
  Arms: Postoperative topical mucopolysaccharide polysulfate cream
Other: Control group — In Control group, only standard therapy was performed after surgery
  Arms: Control group

SUMMARY:
The present study was to evaluate the effect of topical Arnica and MPSP application with respect to visual analogue scale (VAS) scores, maximal interincisal opening (MIO) and edema values after mandibular impacted third molar removal on days 1, 3, 5 and 10 postoperatively. The following null hypotheses of the present research were determined as follows: usage of topical agents would not influence i) VAS scores, ii) MIO values, and iii) edema values on 1st, 3rd, 5th, and 10th days after the mandibular impacted third molar surgery

ELIGIBILITY:
Inclusion Criteria:

* Age between 16-68 years
* American Society of Anesthesiologists (ASA) Class 1 physiological status
* Consistent radiological and clinical data
* Volunteered to participate in the study
* Scale II" surgery difficulty according to Modified Parant Classification for mandibular impacted third molar removal, be free of pericoronitis and infection at operation time

Exclusion Criteria:

* Being out of age range
* Pregnancy or lactation
* Analgesic or antibiotic therapy history in last 14 days due to symptoms of related third molar
* Smoking cigarette
* Any pathology associated with impacted third molar
* Active complaints on preoperative examination on the day of surgery
* Immunosuppressed or diagnosed with malignancy
* Diagnosed chronic diseases such as; Diabetes mellitus (DM), hypertension, cerebrovascular event, psychiatric diseases, coagulopathies
* Autoimmune diseases
* Patients who could not attend regular follow-up visits
* Allergy to the medications prescribed or utilized in study protocol
* Inconsistent clinical and radiological data or missed follow-up

Ages: 16 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Preoperative Pain Intensity | On the day of surgery preoperatively
  The patients were assessed using a visual analogue scale (VAS), 10 cm in length, ranging from 0 for "no pain" to 10 for "the worst possible pain". Preoperative VAS value recorded.
Change From Baseline Maximal Interincisal Opening (MIO) on Postoperative Follow Up Visits | Preoperatively on the day of surgery, postoperative first, third, fifth and tenth days
  All patients' maximal interincisal opening were measured and recorded as the distance between upper and lower central incisors. Preoperative MIO value recorded. The measurements were repeated as described above in the 1st, 3rd, 5th, and 10th days after surgery and recorded.
3. Change From Baseline Facial Measurements for Evaluation of Edema on Postoperative Follow Up Visits | Preoperatively on the day of surgery, postoperative first, third, fifth and tenth days
  The level of edema was determined by a modification of tape measuring method described by Gabka and Matsumara [20, 21]. Three measurements (in mm) (AC, AE and BE) were made between 5 reference points: A) tragus, B) lateral corner of the eye, C) outer corner of the mouth, D) angle of the mandible, and E) soft tissue pogonion. The mean of three preoperative measurements was calculated and recorded. The measurements were repeated as described above in the 1st, 3rd, 5th, and 10th days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Neşet Akay, Study Director — Abant Izzet Baysal University
Locations (1):
- Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) related to study protocol and results will be shared during submitting as an article.
Supporting Information: Study Protocol
Time Frame: The present study will be transformed to an article in six months
Access Criteria: All IPD and supporting information data will be accessible after publication of the article

REFERENCES:
- [Result] Simsek G, Sari E, Kilic R, Bayar Muluk N. Topical Application of Arnica and Mucopolysaccharide Polysulfate Attenuates Periorbital Edema and Ecchymosis in Open Rhinoplasty: A Randomized Controlled Clinical Study. Plast Reconstr Surg. 2016 Mar;137(3):530e-535e. doi: 10.1097/01.prs.0000479967.94459.1c. PMID 26910697
- [Result] Lokken P, Straumsheim PA, Tveiten D, Skjelbred P, Borchgrevink CF. Effect of homoeopathy on pain and other events after acute trauma: placebo controlled trial with bilateral oral surgery. BMJ. 1995 Jun 3;310(6992):1439-42. doi: 10.1136/bmj.310.6992.1439. PMID 7613277
- [Result] Sindet-Pedersen S, Lund E, Simonsen EK, Stenbjerg S. The anti-inflammatory effect of organo-heparinoid cream after bilateral mandibular osteotomies. Int J Oral Maxillofac Surg. 1989 Feb;18(1):35-8. doi: 10.1016/s0901-5027(89)80013-x. PMID 2469747
- [Derived] Akay N, Sanal KO. Can Topical Agents (Arnica and Mucopolysaccharide Polysulfate) Reduce Postoperative Pain, Edema and Trismus Following Mandibular Third Molar Surgery? J Oral Maxillofac Surg. 2024 Jan;82(1):113-121. doi: 10.1016/j.joms.2023.10.003. Epub 2023 Oct 12. PMID 37913818